CLINICAL TRIAL: NCT01049724
Title: Lacritin and Heparanase Levels in Human Tears After Laser Refractive Surgery
Status: Completed | Type: Observational
Sponsor: Fort Belvoir Community Hospital (U.S. Federal Agency)
Collaborators: James Madison University (Other); University of Virginia (Other)
Responsible Party: Principal Investigator, COL Bruce Rivers, Director, Warfighter Refractive Eye Surgery Program and Research Center at FT Belvoir, Fort Belvoir Community Hospital
Other Study IDs: 351515
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Myopia
Keywords: Myopia; refractive surgery; LASIK; PRK; Lacritin; Heparanase
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- PRK: Those patients undergoing photorefractive keratectomy
  Interventions: Other: Tear collection
- LASIK: Those undergoing Laser-assisted insitu keratomileusis
  Interventions: Other: Tear collection

INTERVENTIONS:
Other: Tear collection — Tear collection

SUMMARY:
The purpose of this study is to measure tear lacritin and heparanase levels before and following surgery using a minimal risk procedure to collect tears from patients undergoing PRK or LASIK.

DETAILED DESCRIPTION:
Lacritin is a naturally occurring tear protein with antimicrobial activity that is capable of stimulating mitogenesis in human corneal epithelial cells and promoting production of tears in lacrimal gland acinar cells. A recently developed immunoassay for lacritin may help characterize the lacritin response following refractive surgery with the possible development of recombinant lacritin as a novel therapeutic agent for wound healing. Heparanase (HPSE) acts as a regulator for lacritin by cleaving heparan sulfate chains and allowing lacritin to bind. We aim to measure both tear lacritin and HPSE pre- and post-operatively to elucidate lacritin and HPSE's response in patients undergoing PRK (photorefractive keratectomy) and LASIK (Laser-assisted in situ keratomileusis) at the Walter Reed Center for Refractive Surgery.

ELIGIBILITY:
Inclusion Criteria:

* Active duty US Army Soldiers eligible for care at FBCH
* Undergoing PRK or LASIK
* Male or female, of any race, and at least 21 years old and not older than 55 years old at the time of the tear collection. The lower age limit of 21 years is intended to ensure documentation of refractive stability.
* Appropriately aged individuals who report that their eyes are "normal" and who have no active eye illness as determined by the principal investigator or sub-investigator.
* Ability and willingness to understand and provide informed consent to participate in this study.
* Up to -10.00 diopters of myopia.
* Subject must expect to be located in the greater Washington DC area for a 12 month period post-operatively.
* Consent of the subject's command (active duty) to participate in the study.
* Access to transportation to meet follow-up requirements.

Exclusion Criteria:

* Any reason to be excluded for PRK or LASIK
* Female subjects who are pregnant, breast-feeding or intend to become pregnant during the study. Female subjects will be given a urine pregnancy test prior to participating in the study to rule out pregnancy. [Pregnancy and breastfeeding are contraindications to refractive surgery in general, including PRK, whether participating in this study or not]
* Patients with known sensitivity or inappropriate responsiveness to any of the medications used in the post-operative course.
* Any physical or mental impairment that would preclude participation in any of the examinations.
* Anterior basement membrane dystrophy
* History of recurrent epithelial erosion
* Significant dry eye (symptomatic with Schirmer <5mm at 5 minutes)
* Other corneal epithelial disorder or healing abnormality
* Individuals with any infectious or inflammatory ocular conditions (e.g. have "pink eye" or uveitis).
* Individuals diagnosed with dry eye or other ocular surface condition, including but not restricted to neurotropic keratitis, anterior basement membrane dystrophy, and recurrent corneal erosions.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Active duty military aged 21 to 55 with myopia up to -10.00 diopters eligible for care at Walter Reed Army Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2010-01; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is tear lacritin levels pre- and post-surgery. | pre and standard visits up to 6 months post-surgery

SECONDARY OUTCOMES:
The secondary outcome is tear heparanase levels pre- and post-surgery | pre- and at standard visits up to 6 months post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kraig S. Bower, MD, Principal Investigator — The Wilmer Eye Institute, Johns Hopkins University
Locations (1):
- Fort Belvoir Community Hospital, Fort Belvoir, Virginia, United States